CLINICAL TRIAL: NCT07403747
Title: Evaluation of the Effects of Ride-On Toy Car Use During Operating Room Transfer on Preoperative Anxiety and Postoperative Delirium in Preschool Children
Brief Title: Ride-On Toy Car Use During Operating Room Transfer in Preschool Children
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Filiz Kaya, M.D., Ankara City Hospital Bilkent
Other Study IDs: TABED 1-25-1794
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Preoperative Anxiety; Emergence Delirium in Pediatric Anesthesia
Keywords: Pediatric anesthesia; Preoperative anxiety; Toy car intervention; Emergence delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Toy Car Transfer: Participants will be transferred to the operating room using a ride-on toy car.
  Interventions: Other: Toy car
- Standard Stretcher Transfer: Participants will be transferred to the operating room using a standard hospital stretcher
  Interventions: Other: Standard Transfer

INTERVENTIONS:
Other: Toy car — Transfer to the operating room using a ride-on toy car.
  Groups: Toy Car Transfer
Other: Standard Transfer — Transfer to the operating room using a standard hospital stretcher.
  Groups: Standard Stretcher Transfer

SUMMARY:
The goal of this clinical trial is to determine whether the method of transfer to the operating room can reduce preoperative anxiety and postoperative emergence delirium in male children aged 3 to 7 years undergoing elective adenoidectomy and/or tonsillectomy.

The main questions it aims to answer are:

* Does transfer using a ride-on toy car reduce preoperative anxiety compared with standard stretcher transfer?
* Does this transfer method affect the incidence and severity of postoperative emergence delirium? Researchers will compare toy car transfer with standard hospital stretcher transfer to see if the toy car transfer is associated with lower anxiety levels and reduced emergence delirium.

Participants will:

* Transfer to the operating room either using a ride-on toy car or a standard hospital stretcher
* Have preoperative anxiety assessed at predefined time points
* Be evaluated for postoperative emergence delirium during recovery

DETAILED DESCRIPTION:
This study is designed to investigate the effect of the method of transfer to the operating room on preoperative anxiety levels and postoperative emergence delirium in pediatric patients. This study is designed to investigate the effect of the method of transfer to the operating room on preoperative anxiety levels and postoperative emergence delirium in pediatric patients. The study will include male children aged 3 to 7 years who are scheduled for elective adenoidectomy and/or tonsillectomy under general anesthesia.

Participants will be allocated into two groups. In Group 1, children will be transferred from the waiting area to the operating room using a ride-on toy car. In Group 2, children will be transferred using a standard hospital stretcher according to routine clinical practice. All other perioperative anesthesia management protocols will be standardized between groups.

Preoperative anxiety will be assessed at four predefined time points: in the waiting area (T0), immediately before transfer to the operating room (T1), in the operating room corridor (T2), and immediately before anesthesia induction (T3). Anxiety levels will be measured using the Modified Yale Preoperative Anxiety Scale (m-YPAS) and the Visual Analog Scale for Anxiety (VAS-A).

Postoperative emergence delirium will be evaluated using the Pediatric Anesthesia Emergence Delirium (PAED) scale at three time points: immediately after extubation (P0), upon admission to the post-anesthesia care unit (P1), and 30 minutes after admission to the post-anesthesia care unit (P2).

The primary outcome of the study is the difference in preoperative anxiety levels between the two groups. Secondary outcomes include the incidence and severity of postoperative emergence delirium. The findings of this study may contribute to the development of simple, non-pharmacological strategies to improve perioperative psychological well-being and postoperative recovery in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Male children aged 3 to 7 years scheduled for elective adenoidectomy and/or tonsillectomy under general anesthesia
* Ability to communicate verbally
* American Society of Anesthesiologists (ASA) physical status I or II
* Written informed consent obtained from a parent or legal guardian

Exclusion Criteria:

* Presence of psychiatric disorders, genetic diseases, neurological or developmental disorders
* Chronic pain conditions or ongoing medical treatments that may affect anxiety levels
* Refusal to participate despite repeated encouragement by the investigators
* Use of additional anxiolytic interventions or medications prior to the intervention outside the study protocol
* Previous history of surgical procedures

Ages: 3 Years to 7 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Study Population: Male pediatric patients aged 3 to 7 years scheduled for elective adenoidectomy and/or tonsillectomy under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Preoperative Anxiety Level | Assessments will be conducted in the waiting area, immediately before transfer to the operating room, during transport through the operating room corridor, and immediately before anesthesia induction.
  Preoperative anxiety will be assessed using the Modified Yale Preoperative Anxiety Scale (m-YPAS) and the Visual Analog Scale for Anxiety (VAS-A) during the preoperative period. Preoperative anxiety will be assessed using m-YPAS, (score range 23-100) and VAS-A (score range 0-10), with higher scores indicating increased anxiety severity.

SECONDARY OUTCOMES:
Postoperative Emergence Delirium | From extubation through 30 minutes after admission to the post-anesthesia care unit
  Emergence delirium will be assessed using the Pediatric Anesthesia Emergence Delirium Scale (PAED; total score range 0-20). A score ≥10 will be considered indicative of emergence delirium, with higher scores reflecting greater severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data including demographic characteristics, group assignment, preoperative anxiety scores, and postoperative emergence delirium scores will be shared.
Supporting Information: Study Protocol
Time Frame: Beginning after publication of the primary results and continuing indefinitely.
Access Criteria: De-identified individual participant data and the study protocol will be shared with qualified researchers upon reasonable request and approval by the principal investigator.

REFERENCES:
- [Background] Vakili R, Feizi R, Salimi Y, Mottahedi M, Rizevandi P. Play dough or balloon blowing? A clinical trial comparing creative interventions for reducing preoperative anxiety in children aged 4-8 years. BMC Pediatr. 2025 May 15;25(1):384. doi: 10.1186/s12887-025-05718-1. PMID 40375092
- [Background] Iarikov DE, Shevelev IN, Baskov AV. [International standards in assessing the neurological disorders in spinal and spinal cord trauma]. Zh Vopr Neirokhir Im N N Burdenko. 1999 Jan-Mar;(1):36-8. No abstract available. Russian. PMID 10335578
- [Background] Park SH, Park S, Lee S, Choi JI, Bae HB, You Y, Jeong S. Effect of transportation method on preoperative anxiety in children: a randomized controlled trial. Korean J Anesthesiol. 2020 Feb;73(1):51-57. doi: 10.4097/kja.19191. Epub 2019 Jul 15. PMID 31304694
- [Background] Pastene B, Piclet J, Praud C, Garcia K, Louis K, Schmidt C, Boyadjiev I, Boucekine M, Baumstarck K, Bezulier K, Bouvet L, Zieleskiewicz L, Leone M. Pre-operative distraction using electric ride-on cars for children undergoing elective ambulatory surgery: A randomised controlled trial. Eur J Anaesthesiol. 2023 Mar 1;40(3):190-197. doi: 10.1097/EJA.0000000000001758. Epub 2022 Oct 3. PMID 36204923

DOCUMENTS (1):
  • Study Protocol (2025-10-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT07403747/Prot_000.pdf